CLINICAL TRIAL: NCT07297498
Title: The Effect of Simulation-based Education Within the Framework of the Clinical Judgment Model on Nursing Students' Clinical Decision-making Skills and Perceptions of Nursing Process Competence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, EBRU TURHAL, Lect. Dr., Karadeniz Technical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: E-13562490-050.01.04-620465
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Nursing Process; Clinical Decision Making; Simulation Edication
Keywords: simulation; nursing process; clinical decision making

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulation-Based Training Group (Experimental): Nursing students will receive simulation-based training structured within the Clinical Judgment Model. The intervention aims to improve clinical skills and nursing process competencies. Participants will undergo pre-test measurements before the training session and post-test evaluations after the training.
  Interventions: Other: Siimulation education

INTERVENTIONS:
Other: Siimulation education — Simulation training provided within the framework of the clinical judgment model

SUMMARY:
The purpose of this study is to examine the effects of simulation training delivered within the framework of the clinical judgment model on nursing students' clinical decision-making skills and perceptions of nursing process competency. The research hypothesis is H1: Simulation training delivered within the framework of the clinical judgment model affects nursing students' clinical decision-making skills. H2: Simulation training delivered within the framework of the clinical judgment model affects nursing students' perceptions of nursing process competency.

This study has a single-group pretest-posttest quasi-experimental design. The research population will consist of third-year nursing students in the nursing department at a university located in northern Turkey. The sample will be selected using a convenience sampling method. Participants will first undergo a pretest and then participate in simulation-based training delivered within the framework of the clinical judgment model. A posttest will then be administered.

ELIGIBILITY:
Inclusion

* Criteria:not having had any previous simulation training experience
* Being a 3rd year nursing student
* volunteering to participate in the study

Exclusion Criteria:

* have previous experience with simulation-based training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
clinical decision-making skills | 8 week
  Students' clinical decision-making skills will be measured using the Nursing Clinical Decision-Making Scale and the Lasater Clinical Judgment Rubric.
perception of competence in the nursing process | 8 week
  Nursing process competency perception of students before and after the training will be evaluated with the nursing process competency scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared